CLINICAL TRIAL: NCT00639691
Title: A Compassionate Access Protocol to Assess the Safety of XolairTM (Omalizumab)in Patients (≥ 6 Years Old) With Severe Allergic Asthma Who Remain Symptomatic Despite Optimal Therapy
Brief Title: A Compassionate Access Protocol to Assess the Safety of XolairTM (Omalizumab) in Patients (≥ 6 Years Old) With Severe Allergic Asthma Who Remain Symptomatic Despite Optimal Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025ACA01
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma, Anti-immunoglobin E, omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: omalizumab

INTERVENTIONS:
Biological: omalizumab — sc

SUMMARY:
This study has the objective of providing compassionate use access to omalizumab (Xolair) and to evaluate the Safety of Xolair in subjects with severe allergic asthma who remain symptomatic despite optimal therapy according to GINA step 4 treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* male or female, ≥ 6years of age;
* who have a diagnosis of allergic asthma ≥ 1 year duration according to American Thoracic Society (ATS) criteria;
* severe persistent allergic asthma who remain symptomatic despite optimal therapy (as per Canadian Asthma Consensus Report (1999));
* Subjects having successfully completed one of the following protocols: CIGE025A011E3, CIGE025A2425, CIGE025AIA05;
* elevated immunoglobin E levels

Exclusion Criteria:

* significant systemic disease
* pregnancy or lactation
* an active lung disease other than allergic asthma (eg: cystic fibrosis, bronchiestasis);
* history of food or drug related severe anaphylactoid or anaphylactic reaction(s);
* current treatment with warfarin (Coumadin®), immunomodulatory therapy (e.g., methotrexate, gold, cyclosporine), or antiplatelet therapy.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events from first visit until end of study

SECONDARY OUTCOMES:
To evaluate reasons for premature discontinuation.
All adverse events, duration of study participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Montreal, Quebec, Canada